CLINICAL TRIAL: NCT02629913
Title: Is Internet-based Self-help Effective for the Treatment of Insomnia Disorder?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mementor somnium
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Waiting Lists

ARMS (2):
- Intervention (Experimental): mementor somnium
  Interventions: Device: mementor somnium
- Waitlist (Other)
  Interventions: Other: wait list

INTERVENTIONS:
Device: mementor somnium
  Arms: Intervention
Other: wait list — delayed access to mementor somnium
  Arms: Waitlist

SUMMARY:
The Swiss company mementor has recently developed an interactive self-help intervention for the treatment of insomnia entitled mementor somnium. This programme is based on the guidelines for cognitive-behavioural therapy. mementor somnium consists of 6 online sessions. An animated personal sleep coach provides relevant audio-information and asks questions to which the patient is invited to respond. The components of the programme flexibly adapt to the patient's responses. Aside from psycho-education, exercises and an instruction for sleep restriction, mementor somnium includes a cognitive restructuring intervention in terms of a Socratic dialogue. This Socratic dialogue, implemented by the animated sleep coach, is based on a complex algorithm in the shape of an decision tree. University of Zurich's Department of Psychology in Switzerland will test the effectiveness of mementor somnium in a randomised controlled trial with three assessment times (pre, 6-weeks post and 3-months follow-up). Patients suffering from insomnia will be allocated randomly to either the active intervention group or the waitlist control group. Participants will have access to the programme mementor somnium for six weeks. Primary outcome measure is the Insomnia Severity Index, secondary outcome measures are Beck Depressions-Inventory revised (BDI-II), Brief Symptom Inventory 18, and the SF-12 Health Survey. Additionally, sleep diary data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia Disorder (DSM-5)
* German language comprehension
* Internet-access

Exclusion Criteria:

* Other sleep disorder
* Suicidality
* Current psychotherapy
* Drug abuse or recent change in medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Six weeks

SECONDARY OUTCOMES:
Beck Depression Inventory | Six weeks
Brief Symptom Inventory 18 | Six weeks
SF-12 Health Survey | Six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland